CLINICAL TRIAL: NCT01428427
Title: A Phase IB Combination Study of MEK Inhibitor GSK1120212 With Gemcitabine in Subjects With Solid Tumors
Brief Title: Combination Study of GSK1120212 With Gemcitabine in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112111
Record Dates: First submitted 2009-12-10; First posted 2011-09-05 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Leukaemia, Myelocytic, Acute
Keywords: Gemcitabine; MEK inhibitor; GSK1120212
MeSH Terms: conditions — Leukemia | interventions — trametinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental): Dose escalation to maximum tolerated dose of GSK1120212 and Gemcitabine.
  Interventions: Drug: GSK1120212; Drug: Gemcitabine

INTERVENTIONS:
Drug: GSK1120212 — Continuous daily oral dosing while on study or disease progression (cycle = 28 days).
Drug: Gemcitabine — Dosing once weekly for 3 weeks in a 28 day cycle until disease progression.

SUMMARY:
MEK112111 is a dose-escalation, Phase IB, open-label, single-arm, multi-center study. The primary objective of the study is to determine the recommended dose and regimen for the orally administered MEK inhibitor GSK1120212 dosed in combination with gemcitabine in subjects with solid tumors.

DETAILED DESCRIPTION:
Subjects will be enrolled using a dose-escalation procedure in which the initial cohort receives a fraction of the GSK1120212 dose that achieved a dose limiting toxicity in a previous study and the recommended dose of gemcitabine. Escalation will proceed until the maximum tolerated doses are identified. These doses will be selected based on emerging safety data. Confirmation of the tolerability of the Recommended Phase II Dose (RP2D) will be explored in approximately 12 subjects. Subjects will continue on treatment until treatment discontinuation criteria are met (disease progression, intercurrent illness, adverse event or consent withdrawal).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Age 18 years old or older and able to swallow oral medication.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology (ECOG) scale.
* Histologically or cytologically confirmed diagnosis of a solid tumor malignancy that is either relapsed or refractory, or potentially responsive to gemcitabine.
* Tumor Type criteria as listed in protocol.
* Male subjects must agree to use one of the contraception methods listed in protocol.
* A female subject is eligible to participate if she is of non-childbearing potential as defined in the protocol or postmenopausal as defined in the protocol. If of child-bearing potential, she agrees to use protocol specified contraceptive methods
* Adequate organ system function as defined below in the protocol.

Exclusion Criteria:

* Chemotherapy, radiotherapy, or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of GSK1120212.
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter preceding the first dose of GSK1120212 - as long as a minimum of 14 days has passed between the last dose of the prior investigational anti-cancer drug and the first dose of GSK1120212.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, dimethy sulfoxide (DMSO), or excipients (See protocol)
* Use of a prohibited medication (as defined in protocol) or current use of anticoagulants (e.g. warfarin, heparin, low molecular weight heparin) at therapeutic levels. Low dose (prophylactic) anticoagulants are permitted provided that subject's prothrombin time (PT) and partial thromboplastin time (PTT) meet entry criteria.
* Gastrointestinal disease predicted to interfere with absorption of an oral drug.
* History of retinal vein occlusion (RVO) or central serous retinopathy.
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein thrombosis.
* Glaucoma diagnosed within one month prior to study day 1.
* Intraocular pressure > 21mm Hg as measured by tonography.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Subjects previously treated for these conditions that are asymptomatic and off corticosteroids for at least two months are permitted. Subjects are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs).
* Unresolved toxicity greater than common terminology criteria for adverse events (CTCAE v4.0) grade 1 from previous anti-cancer therapy.
* History of acute coronary within the past 24 weeks.
* QTc interval greater than or equal to 480 mili seconds (msecs).
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Pregnant or lactating female.
* History of hepatitis B or C. NOTE: Subjects with evidence of cleared hepatitis B infection are permitted [Hepatitis B Surface Antigen (HBsAg) negative, anti-HBsAg positive and anti Hepatitis B core antigen (HBc) positive.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08-12 (Actual); Primary Completion 2011-07-18 (Actual); Study Completion 2011-07-18 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and changes in laboratory values and vital signs. | From date of randomization until withdrawal from the study due to disease progression, AE, withdrawal of consent or study closure approximately 6 months after last subject was randomized.

SECONDARY OUTCOMES:
Tumor response as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v 1.1 | At screening and every 8 weeks until withdrawal from the study due to disease progression, AE, withdrawal of consent or study closure approximately 6 months after last subject was randomized.
drug levels in blood | first 15 days on study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas

REFERENCES:
- [Background] Infante JR, Papadopoulos KP, Bendell JC, Patnaik A, Burris HA 3rd, Rasco D, Jones SF, Smith L, Cox DS, Durante M, Bellew KM, Park JJ, Le NT, Tolcher AW. A phase 1b study of trametinib, an oral Mitogen-activated protein kinase kinase (MEK) inhibitor, in combination with gemcitabine in advanced solid tumours. Eur J Cancer. 2013 Jun;49(9):2077-85. doi: 10.1016/j.ejca.2013.03.020. Epub 2013 Apr 11. PMID 23583440
- See also: Results for study 112111 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112111?search=study&search_terms=112111#rs